CLINICAL TRIAL: NCT04248842
Title: Wireless Assessment of Respiratory and Circulatory Distress in Chronic Obstructive Pulmonary Disease - Validation Study
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Mikkel Elvekjaer, MD, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: WARD-COPD_validation
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Continuous monitoring; Wireless monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous monitoring system — Patients recruited will be continuously monitored with Isansys Lifetouch patch, Isansys wireless blood pressure monitor (Meditech Blue BP-05), Nonin WristOx 3150 as well as departments standard monitors

SUMMARY:
For patients admitted to the medical ward, it is often difficult to predict if their clinical condition will deteriorate, however subtle changes in vital signs are usually present 8 to 24 hours before a life-threatening event such as respiratory failure leading to ICU admission, or unanticipated cardiac arrest. Such adverse trends in clinical observations can be missed, misinterpreted or not appreciated as urgent. New continuous and wearable 27/7 clinical vital parameter monitoring systems offer a unique possibility to identify clinical deterioration before patients condition progress beyond the point-of-no-return, where adverse events are inevitable. As part of the WARD-COPD project, this validation study aim to assess the accuracy of physiologic parameters derived from standard and wireless patient monitors

ELIGIBILITY:
Inclusion Criteria:

- Adult patients admitted with AECOPD

Exclusion Criteria:

* Patient expected not to cooperate
* Patient allergic to plaster, plastic or silicone
* Patients with pacemaker or implantable cardioverter-defibrillator (ICD) unit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with acute exacerbation of COPD will be included in the study upon arrival to the medical ward.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Comparison of heart rate (beats per minute) measurement with Isansys Lifetouch patch vs standard monitoring (Phillips IntelliVue) | Two hours of monitoring (measurement interval of 15 mins)
  Analysed using a Bland Altman (BA) analysis to measure mean difference and limits of agreement between the two methods. The BA analysis will correct for repeated measures within each subject if required.
Comparison of respiratory rate (breaths per minute) measurement with Isansys Lifetouch patch vs standard monitoring (Phillips IntelliVue) vs direct observation | Two hours of monitoring (measurement interval of 15 mins)
  Analysed using a Bland Altman (BA) analysis to measure mean difference and limits of agreement between the three methods. The BA analysis will correct for repeated measures within each subject if required.
Comparison of pulse rate (beats per minute) measurement with Nonin WristOx 3150 vs standard monitoring (Phillips IntelliVue) | Two hours of monitoring (measurement interval of 15 mins)
  Analysed using a Bland Altman (BA) analysis to measure mean difference and limits of agreement between the two methods. The BA analysis will correct for repeated measures within each subject if required.
Comparison of peripheral oxygen saturation (percent) measurement with Nonin WristOx 3150 vs standard monitoring (Phillips IntelliVue) | Two hours of monitoring (measurement interval of 15 mins)
  Analysed using a Bland Altman (BA) analysis to measure mean difference and limits of agreement between the two methods. The BA analysis will correct for repeated measures within each subject if required.
Comparison of systolic and diastolic blood pressure (mmHg) measurement with Meditech BP-05 vs standard monitoring (Phillips IntelliVue) | Two hours of monitoring (measurement interval of 15 mins)
  Analysed using a Bland Altman (BA) analysis to measure mean difference and limits of agreement between the two methods. The BA analysis will correct for repeated measures within each subject if required.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyhoff, MD, PHD, Study Chair — Bispebjerg and Frederiksberg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elvekjaer M, Carlsson CJ, Rasmussen SM, Porsbjerg CM, Gronbaek KK, Haahr-Raunkjaer C, Sorensen HBD, Aasvang EK, Meyhoff CS. Agreement between wireless and standard measurements of vital signs in acute exacerbation of chronic obstructive pulmonary disease: a clinical validation study. Physiol Meas. 2021 Jun 17;42(5). doi: 10.1088/1361-6579/ac010c. PMID 33984846